CLINICAL TRIAL: NCT05813015
Title: Comparison of With and Without Sequential Single Drug Therapy of S-1 After Adjuvant Chemotherapy With Docetaxel Plus S-1 in Stage III Gastric Cancer
Brief Title: Study of Comparing of With and Without Sequential Therapy of S-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian Chen, head of Gastrointestinal department of second affiliated hospital of Zhejiang University, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZRWC_GC_C001
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced Gastric Adenocarcinoma; Chemotherapy Effect
MeSH Terms: interventions — Docetaxel; tegafur-gimeracil-oteracil; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-S group (Experimental): All patients pathologically confirmed pTNM stage III, will receive 6 cycles of DS chemotherapy, and sequential S-1 chemotherapy till 1 year postoperation.
  Interventions: Drug: Docetaxel; Drug: Tegafur-Gimeracil-Oteracil

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 40mg/m2，every 21 days，6 cycles.
Drug: Tegafur-Gimeracil-Oteracil — S-1 40-60mg/m2，p.o, BID, day 1-14, till 1 year postoperation.
  Other Names: S-1

SUMMARY:
The goal of this single arm clinical trial is to learn about sequential S-1 adjuvant therapy in patient wich locally advanced gastric cancer. The main question it aims to answer is:

• The efficacy and safety of S-1 adjuvant therapy, following D2 radical surgery and DS(Docetaxel + S-1) adjuvant chemotherapy.

All patients with locally advanced gastric cancer will received D2 radical surgery, 6 cycles of DS chemotherapy, and sequential S-1 chemotherapy up to 1 year postoperation.

ELIGIBILITY:
Inclusion Criteria:

* (1) Histologically or cytologically confirmed adenocarcinoma of the stomach or adenocarcinoma of the gastroesophageal junction;
* (2) Radical surgery (D2 lymph node dissection) for gastric cancer in our center, with postoperative pathological stage of stage III;
* (3) No significant tumor recurrence or metastasis as assessed by imaging;
* (4) Age 18 years - 75 years;
* (5) ECOG score of 0 or 1;
* (6) Laboratory tests tolerant to chemotherapy;
* (7) Hematological examination: no obvious signs of hematologic diseases, ANC ≥ 1.5 × 10^9/L, platelet count ≥ 80 × 10^9/L, Hb ≥ 90 g/L, WBC ≥ 3.0 × 10^9/L before enrollment, and no bleeding tendency; (8) Biochemical examination: total bilirubin < 1.5 times the upper limit of normal value, AST, ALT < 2.5 times the upper limit of normal value, creatinine < 1.5 times the upper limit of normal value.

Exclusion Criteria:

* (1) Other pathological types of tumors;
* (2) Pregnant or nursing women;
* (3) Those with a history of other malignant neoplastic disease in the last 5 years;
* (4) Those with a history of uncontrolled epilepsy, central nervous system disease, or psychiatric disorder, where the investigator determines whether the clinical severity prevents signing an informed consent form or affects the patient's compliance with oral medications;
* (5) Clinically severe (i.e., active) heart disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or arrhythmias requiring pharmacologic intervention, or a history of myocardial infarction within the last 12 months;
* (6) Severe diabetes-related complications, such as diabetic nephropathy, diabetic ketosis, etc;
* (7) Those with digestive tract obstruction or physiological abnormalities, or suffering from malabsorption syndrome, which may affect S-1 absorption;
* (8) Those who have had gastrointestinal bleeding in the last two weeks, or are at high risk of bleeding as judged by the investigator;
* (9) Known to have peripheral nerve disease ≥ NCI-CTC AE grade 1. but with deep tendon reflexes (DTR) only;
* (10) Those requiring immunosuppressive therapy for organ transplantation;
* (11) who have received other chemotherapy regimens
* (12) Those with uncontrolled severe infections, or other serious concomitant diseases;
* (13) Allergic to S-1 or any of the study drug components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | 3 years
  Recurrence free survival

SECONDARY OUTCOMES:
Overall survival | up to 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal Department of Second Affiliated Hospital of Zhejiang University, Hanzhou, Zhejiang, China